CLINICAL TRIAL: NCT02518243
Title: Safe & Easy for Alzheimer's Disease and Related Pathologies
Acronym: SaFEE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-PP-08
Record Dates: First submitted 2015-07-07; First posted 2015-08-07 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cognitive Deterioration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alzheimer's Disease (Experimental)
  Interventions: Other: Patient's answer with non pharmacological therapeutic

INTERVENTIONS:
Other: Patient's answer with non pharmacological therapeutic — Installation at patient's home of :
  * aromatherapy
  * music therapy
  * cognitive training in multimedia application offering cognitive games

SUMMARY:
All over the world the increasing prevalence of chronic disorders and its impact on functional decline is challenging the sustainability of health care systems. Older individuals also frequently experience the reversible "frailty syndrome", which overlaps with chronic diseases, increasing incidence of disability.

Building a global system aiming to take in charge all causes leading to loss of autonomy is a rather complicated task involving numerous Information and Communication technologies (ICT) solutions which are not always easy to use in everyday life.

The SafEE (Safe Easy Environment) project aim is to improve the safety, autonomy and quality of life of older people at risk.

The SafEE2 project develop non pharmacological therapeutic through diferent ICT (stimulation aromatherapy automatic fragrance ...) .

The goal of this study is to validate the acceptability, sensitivity and efficacy of the systems.

DETAILED DESCRIPTION:
The non pharmacological therapeutic will be install at hospital room :

* aromatherapy,
* music therapy,
* cognitive training in multimedia application offering cognitive games.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of Alzheimer's disease according to NINCDS-ADRDA (McKhann, Drachman et al. 1984) or typical or atypical Alzheimer's disease (Dubois B. et al. 2007).
* Score at Mini Mental Test (MMSE) ≥16.
* Subjects residing in nursing homes.
* Subjects beneficiaries of a social security scheme.
* Signature of free and informed consent.

Exclusion Criteria:

* Failure to pass the neuropsychological tests because of a sensory or motor deficit.
* Sensory deficit (olfactory or visual) preventing the patient made perfectly meet the therapeutic solutions.
* Prescription of a new treatment psychotropic (hypnotic, anxiolytic, antidepressant, antipsychotic) in the week before the evaluation;
* Persons deprived of liberty (administrative or judicial).

Ages: 60 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Tolerance of the systems set up and use frequency evaluated using the Caregiver Questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Renaud DAVID, MD, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- Ehpad Valrose, Nice, France